CLINICAL TRIAL: NCT04289831
Title: "Impact of Preoperative Biliary Drainage on Surgical and Oncologic Outcomes After Pancreatico-Duodenectomy in Patients With Operable Malignant Periampulary Tumors. A Randomized Controlled Study"
Brief Title: Preoperative Biliary Drainage in Patients With Operable Malignant Periampulary Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alexandria (Other)
Responsible Party: Principal Investigator, Mohamed El Messiry, Ass. Professor, University of Alexandria
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 03027612
Record Dates: First submitted 2020-02-27; First posted 2020-02-28 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Periampullary Cancer; Biliary Obstruction; Preoperative Biliary Drainage
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Direct Surgery (DS) group (Active Comparator): patients subjected to direct surgery (DS) within 1 week after randomization
  Interventions: Procedure: Surgery
- Preoperative Biliary Drainage (PBD) group (Active Comparator): patients managed by Preoperative Biliary Drainage followed by surgery after 4-6 weeks.
  Interventions: Procedure: Preoperative Biliary Drainage (PBD); Procedure: Surgery

INTERVENTIONS:
Procedure: Preoperative Biliary Drainage (PBD) — Endoscopic retrograde biliary drainage (ERBD) and stent placement was the first choice for PBD while ultrasound-guided percutaneous transhepatic biliary drainage (PTBD) was done if ERBD was not feasible. Biliary drainage was considered successful if the serum bilirubin level decreased by 50% or more within 2 weeks after the procedure. Patients with failed PBD were referred directly to surgery, while those with successful PBD were referred to surgery 4 to 6 weeks after first drainage procedure according to the latest guidelines
  Arms: Preoperative Biliary Drainage (PBD) group
Procedure: Surgery — The standard surgical procedure for operable tumors Whipple procedure with triple reconstruction, namely pancreatogastrostomy or pancreatojejunostomy,hepaticojejunostomy and gastrojejunostomy

SUMMARY:
The impact of preoperative biliary drainage (PBD) on morbidity and mortality associated with Pancreaticoduodenectomy (PD) in patients with peri-ampulary tumors is still controversial. The objective of this study is to evaluate the impact of PBD on surgical and oncologic outcomes after PD in jaundiced patients with operable peri-ampulary tumors.

DETAILED DESCRIPTION:
150 consecutive jaundiced patients with suspected operable peri-ampullary tumors were randomized via concealed envelopes into 2 groups (each included 75 patients), group I managed by direct surgery while group II managed by PBD followed by surgery. Both groups were compared regarding perioperative mortality, morbidities, tumor recurrence and 2 years survival rates.

ELIGIBILITY:
Inclusion Criteria:

* Serum bilirubin level above 4 mg/dl
* suspected peri-ampullary tumor at computed tomography (CT)
* No evidence of distant metastasis or locally advanced tumor

Exclusion Criteria:

* Patients with evidence of distant metastasis or locally advanced tumor
* Prior neoadjuvant chemotherapy or Radiotherapy
* Prior biliary surgery
* Patients with contraindication for major surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Early postoperative mortality (within 3 months) | within 90 days after surgery
  Death within 90 days postoperatively
Early postoperative morbidities (within 3 months) | within 90 days after surgery
  Any complications related to surgery within 3 months including: postoperative bleeding, pancreatic fistula, Biliary leakage, Intra-abdominal infection, wound infection/ dehiscence

SECONDARY OUTCOMES:
Tumor recurrence | 2 years follow up after surgery
  Local or systemic recurrence of the malignant tumor
Disease free survival (DFS) | 2 years follow up after surgery
  % of patients survived without any evidence of tumor recurrence after 2 years follow up
Overall survival (OS) | 2 years follow up after surgery
  % of patients survived with or without tumor recurrence after 2 years follow up

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed M Elmessiry, MD,PhD, Principal Investigator — Ass. Professor of Surgery (Surgical Oncology Unit); Eman A Mohamed, MD, PhD, Principal Investigator — Lecturer of Internal Medicine (Gastroenterology Unit)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang C, Xu Y, Lu X. Should preoperative biliary drainage be routinely performed for obstructive jaundice with resectable tumor? Hepatobiliary Surg Nutr. 2013 Oct;2(5):266-71. doi: 10.3978/j.issn.2304-3881.2013.09.01. PMID 24570957
- [Background] Mezhir JJ, Brennan MF, Baser RE, D'Angelica MI, Fong Y, DeMatteo RP, Jarnagin WR, Allen PJ. A matched case-control study of preoperative biliary drainage in patients with pancreatic adenocarcinoma: routine drainage is not justified. J Gastrointest Surg. 2009 Dec;13(12):2163-9. doi: 10.1007/s11605-009-1046-9. Epub 2009 Sep 23. PMID 19774424
- [Background] Smith RA, Dajani K, Dodd S, Whelan P, Raraty M, Sutton R, Campbell F, Neoptolemos JP, Ghaneh P. Preoperative resolution of jaundice following biliary stenting predicts more favourable early survival in resected pancreatic ductal adenocarcinoma. Ann Surg Oncol. 2008 Nov;15(11):3138-46. doi: 10.1245/s10434-008-0148-z. Epub 2008 Sep 12. PMID 18787902
- [Background] Abdullah SA, Gupta T, Jaafar KA, Chung YF, Ooi LL, Mesenas SJ. Ampullary carcinoma: effect of preoperative biliary drainage on surgical outcome. World J Gastroenterol. 2009 Jun 21;15(23):2908-12. doi: 10.3748/wjg.15.2908. PMID 19533815